CLINICAL TRIAL: NCT01279161
Title: The Role of FTO Gene Polymorphism and Insulin Preparation in Overweight/Obesity in Children With Type 1 Diabetes Mellitus
Brief Title: The Role of FTO Gene Polymorphism and Insulin Preparation in Obesity in Children With Type 1 Diabetes Mellitus
Acronym: FTO_T1DM
Status: Completed | Type: Observational
Sponsor: University of Bialystok (Other Government)
Responsible Party: Principal Investigator, Wlodzimierz Luczynski, Professor, University of Bialystok
Other Study IDs: FTO DIAB
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: overweight, obesity, children, insulin, pump therapy, FTO
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Small amount of peripheral blood for isolation of DNA for assessment of FTO polymorphism.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- diabetes: The study will include 1500 children with type 1 diabetes, aged 6-18 years. These will be patients from Diabetes Outpatient Clinics and patients hospitalized in Departments of Paediatrics, Endocrinology and Diabetology in University and Municipal Hospitals from Poland (Białystok, Warszawa, Łódź, Gdańsk, Wrocław, Katowice).
- control: Reference group will be made of 1500 children from the above mentioned Clinics and Departments in whom type 1 diabetes was excluded. In these children diagnostics procedures will be conducted for reasons other than body weigh related diseases (excluding simple obesity). The children will not receive any treatment that might influence their body weight.

SUMMARY:
The project aims at assessment of the effect of the FTO gene polymorphism and the type of treatment on the development of overweight/obesity and features of metabolic syndrome in children with type 1 diabetes.

Gene polymorphism including some genetic variants may predispose to the development of cardiovascular diseases and their complications. The A allele of the FTO gene predisposing to obesity occurs in approximately 40% of the European population and each copy of this allele can increase BMI by 0.1 Z-score i.e. by 0.4 kg/m2. Insulin therapy in diabetic patients may result in excess body weight gain. Therefore we need studies involving large groups of children and assessing cardiovascular risk factors in type 1 diabetes along with their genetic associations.

Patients: The study will include 1500 children with type 1 diabetes, aged 6-18 years. Reference group will be made of 1500 children in whom type 1 diabetes was excluded. The following variables will be assessed in the treatment group: 1) Anthropometric data and questionnaire data: age, sex, body height and weight, body mass index (BMI), waist and hip circumferences, arm and thigh circumferences, family history of overweight/obesity, type 1 or 2 diabetes or cardiovascular disease, 2) Primary disease characteristics: age of the disease onset, treatment regimen, mean daily insulin consumption per kg body weight, brands of insulin products, glycated haemoglobin, BMI from the first 3-6 months following diabetes onset, diet, conversion of these data into actual and ideal calorie intake 3) Laboratory data - lipid profile and blood pressure (average of three measurements). Methodology: Gene polymorphism analysis in the extracted DNA will be made with the real-time PCR method using TaqMan 7900 HT by Applied Biosystems. Correlations between the FTO gene polymorphism and clinical variables such as BMI (including BMI increase since the disease onset), body weight and height, waist and hip circumferences, arm and thigh circumferences, and blood pressure will be assessed by a professional statistician with a specially dedicated software. Moreover parameters such as diet and metabolic control will be assessed. As regards insulin therapy the following variables will be analysed: insulin injection device, therapy regimen (intensive versus functional; brands and types of insulin products: human insulin versus insulin analogue), consumption of insulin. All of the above listed variables will be correlated with the genotypes found in the gene polymorphism analysis. The study has been approved by Bioethics Committee of the Medical University in Białystok.

Results: The authors of the project expect that the effect of the FTO gene polymorphism on overweight/obesity and features of metabolic syndrome in children with type 1 diabetes will be shown. Moreover the project will enable assessment of the effect of the therapeutic regimen, including the type of insulin product, on body weight increase in the course of type 1 diabetes treatment in the context of the FTO gene polymorphism. Confirmation of the above associations and identification of a group at risk of excess body weight increase in the course of insulin therapy may help physicians, parents and patients to avoid this complication. Therefore clinical benefit of this project will include identification - based on the genetic assays results - of a group of type 1 diabetic children particularly likely to develop overweight, obesity and other cardiovascular risk factors.

DETAILED DESCRIPTION:
Aim:

The project aims at assessment of the effect of the FTO gene polymorphism and the type of treatment on the development of overweight/obesity and features of metabolic syndrome in children with type 1 diabetes. Particular objective of the project is providing an answer to the question: Are type 1 diabetic children who are carriers of the AA genotype of the FTO gene polymorphism (rs9939609) at risk of more weight gain in the course of insulin therapy when compared to carriers of the TA and TT genotypes of this polymorphism ? Background: Gene polymorphism including some genetic variants may predispose to the development of cardiovascular diseases and their complications. A great advance in studies on genetic susceptibility to obesity was the discovery of the gene called FTO - fat mass and obesity associated gene. The A allele of the FTO gene predisposing to obesity occurs in approximately 40% of the European population and each copy of this allele can increase BMI by 0.1 Z-score i.e. by 0.4 kg/m2. However, there are very few data on the impact of human genome on body weight change following particular intervention.

An important problem to be dealt with by physicians and type 1 diabetic patients is overweight and obesity. This problem is inevitably associated with insulin therapy and excess energy intake. Insulin therapy in diabetic patients may result in excess body weight gain. The exact mechanisms underlying this phenomenon are not known. Obesity in patients diagnosed with diabetes can be an additional risk factor of cardiovascular disease. Central obesity, insulin resistance, dyslipidaemia and arterial hypertension are all the elements of metabolic syndrome - a disease that predisposes to the development of cardiovascular disorders. Cardiovascular complications are the main cause of morbidity and mortality in adult patients with diabetes. However recently repeated attempts have been made to assess these factors also in children and adolescents. Overweight and obesity in type 1 diabetes depend among others on patients' sex, age and type of treatment. Although the role of gene polymorphism in the development of obesity in adults and children is the subject of extensive investigations, currently there are no reports that would assess genetic aspects of obesity in treatment of type 1 diabetes. Therefore we need studies involving large groups of children and assessing cardiovascular risk factors in type 1 diabetes along with their genetic associations.

Patients: The study will include 1500 children with type 1 diabetes, aged 6-18 years. Reference group will be made of 1500 children in whom type 1 diabetes was excluded.

The following variables will be assessed in the treatment group: 1) Anthropometric data and questionnaire data: age, sex, body height and weight, body mass index (BMI) (including SDS-BMI), waist and hip circumferences, arm and thigh circumferences, family history of overweight/obesity, type 1 or 2 diabetes or cardiovascular disease, 2) Primary disease characteristics: age of the disease onset, treatment regimen (intensive insulin therapy versus functional insulin therapy with a personal insulin pump), mean daily insulin consumption per kg body weight, brands of insulin products, glycated haemoglobin (the last available measurement and the mean value from the last year), BMI from the first 3-6 months following diabetes onset, diet - consumption of carbohydrate and protein-fat exchanges (only in patients using a personal insulin pump), conversion of these data into actual and ideal calorie intake 3) Laboratory data: lipid profile (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides) and blood pressure (average of three measurements). In the control group anthropometric variables and questionnaire data will be assessed along with additional questions.

Methodology: Gene polymorphism analysis in the extracted DNA will be made with the real-time PCR method using TaqMan 7900 HT by Applied Biosystems. Correlations between the FTO gene polymorphism and clinical variables such as BMI (including BMI increase since the disease onset), body weight and height, waist and hip circumferences, arm and thigh circumferences, and blood pressure will be assessed by a professional statistician with a specially dedicated software (R-project). Moreover parameters such as diet and metabolic control will be assessed. As regards insulin therapy the following variables will be analysed: insulin injection device, therapy regimen (intensive versus functional; brands and types of insulin products: human insulin versus insulin analogue), consumption of insulin. Out of laboratory data, lipid metabolism parameters will be assessed. All of the above listed variables will be correlated with the genotypes found in the gene polymorphism analysis. The study has been approved by Bioethics Committee of the Medical University in Białystok.

Results: The authors of the project expect that the effect of the FTO gene polymorphism on overweight/obesity and features of metabolic syndrome in children with type 1 diabetes will be shown. Moreover the project will enable assessment of the effect of the therapeutic regimen, including the type of insulin product, on body weight increase in the course of type 1 diabetes treatment in the context of the FTO gene polymorphism. Confirmation of the above associations and identification of a group at risk of excess body weight increase in the course of insulin therapy may help physicians, parents and patients to avoid this complication. Therefore clinical benefit of this project will include identification - based on the genetic assays results - of a group of type 1 diabetic children particularly likely to develop overweight, obesity and other cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* children of Polish origin
* diagnosed with type 1 diabetes (defined according to the ADA 2010)
* treated with insulin therapy for at least 1 year
* aged ≥ 6 < 18 years
* receiving the same treatment regimen for at least one year
* insulin requirement of > 0.5 U/kg/daily

Exclusion Criteria:

* no consent given by parents/guardians
* chromosome disorders
* autoimmune diseases
* coeliac disease (biopsy-proven)
* thyroid hormone disorders (but not the presence of antithyroid antibodies)
* treatment that might influence body weight
* newly diagnosed diabetes (either type 1, 2, 3 or other types of diabetes)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include 1500 children with type 1 diabetes, aged 6-18 years. These will be patients from Diabetes Outpatient Clinics and patients hospitalized in Departments of Paediatrics, Endocrinology and Diabetology in University and Municipal Hospitals from all over Poland (Białystok, Warszawa, Gdańsk, Katowice, Wrocław). Reference group will be made of 1500 children from the above mentioned Clinics and Departments in whom type 1 diabetes was excluded. In these children diagnostics procedures will be conducted for reasons other than body weigh related diseases (excluding simple obesity). The children will not receive any treatment that might influence their body weight.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Identification of the effect of the FTO gene polymorphism on the development of overweight/obesity in insulin treated children | one year

SECONDARY OUTCOMES:
• Identification of the effect of the following factors: sex, age, duration of disease, therapy regimen, type of insulin product and degree of metabolic control on the development of overweight/ obesity in insulin treated children | one year
• Identification of the effect of genetic polymorphism of the FTO gene on the incidence of metabolic syndrome features in insulin treated children. | one year
• Identification of the effect of genetic polymorphism of the FTO gene on the incidence of overweight, obesity and metabolic syndrome features in children without diabetes. | one year
• Comparison of frequency distribution of FTO gene polymorphism involved in the pathogenesis of obesity in children with diabetes versus children without diabetes. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Wlodzimierz Luczynski, Ass. Prof., Study Chair — Medical University of Bialystok, Poland; Adam Kretowski, Prof, Principal Investigator — Medical University of Bialystok, Poland
Locations (6):
- Poland (6):
  - Department of Pediatrics, Endocrinology and Diabetology, Medical University, Wroclaw, Lower Silesian Voivodeship
  - Department of Pediatrics, Medical University, Warsaw, Masovian Voivodeship
  - Department of Pediatrics, Endocrinology, Diabetology with Cardiology Division, Medical University, Bialystok, Podlaskie Voivodeship
  - Department of Pediatrics, Hematology, Oncology and Endocrinology, Medical University, Gdansk, Pomeranian Voivodeship
  - Department of Pediatrics, Endocrinology and Diabetology, Medical University, Katowice, Silesian Voivodeship
  - Department of Pediatrics, Oncology, Hematology and Diabetology, Medical University, Lodz, Łódź Voivodeship

REFERENCES:
- [Background] Timpson NJ, Emmett PM, Frayling TM, Rogers I, Hattersley AT, McCarthy MI, Davey Smith G. The fat mass- and obesity-associated locus and dietary intake in children. Am J Clin Nutr. 2008 Oct;88(4):971-8. doi: 10.1093/ajcn/88.4.971. PMID 18842783
- [Background] Frayling TM, Timpson NJ, Weedon MN, Zeggini E, Freathy RM, Lindgren CM, Perry JR, Elliott KS, Lango H, Rayner NW, Shields B, Harries LW, Barrett JC, Ellard S, Groves CJ, Knight B, Patch AM, Ness AR, Ebrahim S, Lawlor DA, Ring SM, Ben-Shlomo Y, Jarvelin MR, Sovio U, Bennett AJ, Melzer D, Ferrucci L, Loos RJ, Barroso I, Wareham NJ, Karpe F, Owen KR, Cardon LR, Walker M, Hitman GA, Palmer CN, Doney AS, Morris AD, Smith GD, Hattersley AT, McCarthy MI. A common variant in the FTO gene is associated with body mass index and predisposes to childhood and adult obesity. Science. 2007 May 11;316(5826):889-94. doi: 10.1126/science.1141634. Epub 2007 Apr 12. PMID 17434869
- [Background] Reinehr T, Holl RW, Roth CL, Wiesel T, Stachow R, Wabitsch M, Andler W; DPV-Wiss Study Group. Insulin resistance in children and adolescents with type 1 diabetes mellitus: relation to obesity. Pediatr Diabetes. 2005 Mar;6(1):5-12. doi: 10.1111/j.1399-543X.2005.00093.x. PMID 15787895
- [Background] Luczynski W, Szypowska A, Glowinska-Olszewska B, Bossowski A. Overweight, obesity and features of metabolic syndrome in children with diabetes treated with insulin pump therapy. Eur J Pediatr. 2011 Jul;170(7):891-8. doi: 10.1007/s00431-010-1372-7. Epub 2010 Dec 8. PMID 21140273
- [Derived] Luczynski W, Fendler W, Ramatowska A, Szypowska A, Szadkowska A, Mlynarski W, Chumiecki M, Jarosz-Chobot P, Chrzanowska J, Noczynska A, Brandt A, Mysliwiec M, Glowinska-Olszewska B, Bernatowicz P, Kowalczuk O, Bossowski A. Polymorphism of the FTO Gene Influences Body Weight in Children with Type 1 Diabetes without Severe Obesity. Int J Endocrinol. 2014;2014:630712. doi: 10.1155/2014/630712. Epub 2014 Aug 19. PMID 25214838